CLINICAL TRIAL: NCT05525039
Title: Dissecting the Therapeutic Mechanism of an Effective Combination Treatment Targeting Neuromuscular Junction Dengeneration and Myosteatosis to Combat Sarcopenia
Brief Title: RCT of Combination Effect of Vibration Treatment and HMB Supplementation on Myosteatosis and NMJ Degeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Professor CHEUNG Wing hoi, Louis, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CREC 2022.233-T
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenia; Connective Tissue Diseases in Old Age; Musculoskeletal Abnormalities
Keywords: Sarcopenia; Vibration; Hydroxymethylbutyrate
MeSH Terms: conditions — Sarcopenia; Musculoskeletal Abnormalities

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either (1) Control, (2) HMB only, (3) VT only or (4) HMB +VT group. All subjects will be given protein supplement to ensure minimal daily protein intake. Subject assigned to VT group will receive VT (35Hz, 0.3g, 20min/day, at least 3 times/week) for 6 months. Subjects assigned to HMB group will take HMB capsules 3g/day for 6 months.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Placebo Comparator): Subjects assigned to Contro Group will not receive VT or HMB. They will receive daily protein supplement for 6 months.
  Interventions: Dietary Supplement: Protein supplement
- HMB only Group (Active Comparator): Subjects assigned to HMB only Group will receive HMB supplement at 3g/day and daily protein supplement for 6 months.
  Interventions: Dietary Supplement: β-hydroxy β-methylbutyrate (HMB) supplement; Dietary Supplement: Protein supplement
- VT only Group (Active Comparator): Subjects assigned to VT only Group will receive VT (0.3g, 35Hz, at least 3 times/week) and daily protein supplement for 6 months
  Interventions: Device: Low-magnitude High-frequency Vibration; Dietary Supplement: Protein supplement
- HMB + VT Group (Experimental): Subjects assigned to HMB + VT Group will receive HMB supplement at 3g/day, VT at least 3 times/week and daily protein supplement for 6 months.
  Interventions: Device: Low-magnitude High-frequency Vibration; Dietary Supplement: β-hydroxy β-methylbutyrate (HMB) supplement; Dietary Supplement: Protein supplement

INTERVENTIONS:
Device: Low-magnitude High-frequency Vibration — 0.3g, 35Hz, 20mins/day, at least 3 times/week
  Other Names: Vibration Treatment
  Arms: HMB + VT Group; VT only Group
Dietary Supplement: β-hydroxy β-methylbutyrate (HMB) supplement — Oral nutritional HMB supplement at 3g/day
  Arms: HMB + VT Group; HMB only Group
Dietary Supplement: Protein supplement — Daily protein supplement intake

SUMMARY:
The investigators' pre-clinical study confirms the positive effects of combined treatment (VT + HMB) on reducing fat-to-lean tissue ratio, intramuscular fat infiltration and increasing muscle strength in sarcopenia animal model. The results showed that fat mass could be decreased by ~32%, while histology Oil Red O staining indicated a decrease of fat by almost 60%; in contrast, lean muscle mass increased by ~14%. On muscle strength, combined treatment increased twitch force, tetanic force and grip strength by ~30-66%. These in vivo results are very encouraging and the investigators should explore its potential in clinical translation. As VT and HMB supplement have been commercially available and their compliance rates are satisfactory, they can be translated to clinical application easily. The investigators' next step is to confirm its clinical efficacy, so that sarcopenia becomes a new indication of VT and HMB. The hypothesis is that combined treatment of VT and HMB can retard the progression of sarcopenia in human, in terms of muscle mass, muscle strength and performance.

DETAILED DESCRIPTION:
In this study, a single-blinded RCT is to investigate the effect of combination treatment of VT and HMB on hand grip, gait speed, muscle mass (DXA) in sarcopenic subjects.

Subjects over age of 65 will be screened by performing SARC-F, handgrip, gait speed and bioelectric impedance assessment (BIA) based on AWGS definition. The participants failed in AWGS algorithm will be invited to join the research. Exclusion criteria are those with (1)pathological bone diseases, (2) chronic inflammatory conditions (e.g. rheumatoid arthritis), (3) neurological problems affecting gait, (4) taking regular supervised exercise training for more than 3 times/week, (5) chair-bound or bed-bound, and (6) malignancy.

Recruited subjects will be randomized to either (1) Control, (2) HMB only, (3) VT only or (4) HMB +VT group. All subjects will be given protein supplement to ensure minimal daily protein intake. Subject assigned to VT group will receive VT (35Hz, 0.3g, 20min/day, at least 3 times/week) for 6 months. Subjects assigned to HMB group will take HMB capsules 3g/day for 6 months. Subjects assigned to HMB+VT group will recieve both VT and HMB supplements for 6 months. The primary outcome is muscle strength showing subjects' functional ability. All primary and secondary outcome assessments for all groups will be performed in the investigators' institute at baseline, 3 months and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 60 years or above
* Subjects failed in AWGS algorithm

  1. skeletal muscle mass by BIA (male at <7.0 kg/m^2, female at <5.7 kg/m^2), and
  2. handgrip strength (male at <28 kg, female at <18kg), and/or
  3. gait speed test (>1m/s)

Exclusion Criteria:

* Subjects with pathological bone diseases
* Subjects with chronic inflammatory condition (e.g. rheumatoid arthritis)
* Subjects with neurological problems
* Subjects receiving regular exercise
* Subjecs who are chair-/bed- bound
* Subjects with malignancy
* Subjects with cardiovascular concern such as with pace-maker in-situ
* Subjects with acute fractures or severe osteoarthritis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Muscle strength-handgrip | 6 months
  Handgrip strength will be measured by a dynamometer on each hand of the subject.
Muscle performance-gait speed | 6 months
  Gait speed will be assessed by a 6-meter-walk test.

SECONDARY OUTCOMES:
Dual energy x-ray absortiometry (DXA) | 6 months
  Whole body muscle mass measurement
Biodex Balance System-LOS | 6 months
  Limits of stability will be recorded to evaluate the dynamic posture stability. Maximum scores will be 100 where the higher scores indicate better performance.
Biodex Balance System-OSI | 6 months
  Posture stability (Overall Stability Index) will be recorded. High scores indicate poorer balancing abillity.
Time-up-and-go test (TUG) | 6 months
  Time will be recorded for participants to rise from a chair, walk 3 meters, turn around, and walk back to the chair then sitting down
36-item Short-Form Health Survey (SF-36) | 6 months
  Health-related quality of life will be assessed by the validated Chinese version of SF-36. Scores range from 0 to 100 where higher scores indicate better health status

CONTACTS AND LOCATIONS:
Overall Officials: Wing Hoi Cheung, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Evangelical Luthera Church Social Service - Hong Kong, Hong Kong
  - The Chinese University of Hong Kong Jockey Club Centre for Osteoporosis Care and Control, Hong Kong
  - The Chinese University of Hong Kong, Department of Orthopaedics and Traumatology, 1/F Li Ka Shing Outpatient Clinic (North), PWH, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung KS, Li CY, Tse YK, Choy TK, Leung PC, Hung VW, Chan SY, Leung AH, Cheung WH. Effects of 18-month low-magnitude high-frequency vibration on fall rate and fracture risks in 710 community elderly--a cluster-randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1785-95. doi: 10.1007/s00198-014-2693-6. Epub 2014 Mar 28. PMID 24676848
- [Background] Wang J, Cui C, Chim YN, Yao H, Shi L, Xu J, Wang J, Wong RMY, Leung KS, Chow SK, Cheung WH. Vibration and beta-hydroxy-beta-methylbutyrate treatment suppresses intramuscular fat infiltration and adipogenic differentiation in sarcopenic mice. J Cachexia Sarcopenia Muscle. 2020 Apr;11(2):564-577. doi: 10.1002/jcsm.12535. Epub 2020 Jan 28. PMID 31994349
- [Background] Deutz NE, Pereira SL, Hays NP, Oliver JS, Edens NK, Evans CM, Wolfe RR. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on lean body mass during 10 days of bed rest in older adults. Clin Nutr. 2013 Oct;32(5):704-12. doi: 10.1016/j.clnu.2013.02.011. Epub 2013 Mar 4. PMID 23514626
- [Background] Cheung WH, Mok HW, Qin L, Sze PC, Lee KM, Leung KS. High-frequency whole-body vibration improves balancing ability in elderly women. Arch Phys Med Rehabil. 2007 Jul;88(7):852-7. doi: 10.1016/j.apmr.2007.03.028. PMID 17601464
- [Background] Zhu LY, Chan R, Kwok T, Cheng KC, Ha A, Woo J. Effects of exercise and nutrition supplementation in community-dwelling older Chinese people with sarcopenia: a randomized controlled trial. Age Ageing. 2019 Mar 1;48(2):220-228. doi: 10.1093/ageing/afy179. PMID 30462162
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Derived] Li MCM, Cheng YK, Cui C, Chow SKH, Wong RMY, Kwok TC, Siu PM, Yang M, Tian M, Rubin C, Welch AA, Qin L, Law SW, Cheung WH. Biophysical and nutritional combination treatment for myosteatosis in patients with sarcopenia: a study protocol for single-blinded randomised controlled trial. BMJ Open. 2024 Jan 4;14(1):e074858. doi: 10.1136/bmjopen-2023-074858. PMID 38176874